CLINICAL TRIAL: NCT05129189
Title: Functional Cure Study of Anti-PD-L1 Antibody ASC22 in Combination With Chidamide
Brief Title: Functional Cure Study of Anti-PD-L1 Antibody ASC22 in Combination With Chidamide in HIV-infected Patients With Antiviral Suppression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Jun Chen, MD, Deputy chief physician, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC22
Record Dates: First submitted 2021-11-15; First posted 2021-11-22 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: Functional cure of HIV， ASC22，PD-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASC22 group (Experimental): ASC22 1mg/kg hypodermic injection Q4W+Chidamide 10mg PO BIW
  Interventions: Drug: ASC22 group

INTERVENTIONS:
Drug: ASC22 group — The trial group received ASC22 1mg/kg hypodermic injection Q4W and Chidamide 10mg PO BIW.

SUMMARY:
In HIV-infected patients, enhanced PD-1 expression of T cells correlates with T cell depletion, as evidenced by reduced virus-specific proliferative capacity and decreased cytokine expression.Targeting PD-L1 drugs to block PD-1/PD-L1 signaling may promote the secretion of antiviral cytokines and achieve HIV clearance.The mechanism of action of ASC22 is to competitively block the binding of PD-1 molecules to PD-L1 through its antigen-binding region with a high affinity for hPD-L1, thereby stimulating an innate or adaptive immune response with sustained T-cell activation.This study was conducted to evaluate whether ASC22 combined with chidamide in HIV-infected patients with antiviral suppression could shrink the viral reservoir.

ELIGIBILITY:
Inclusion Criteria:

1. People diagnosed with HIV infection.
2. Age ≥18 years.
3. In good general health with a body mass index ≥18.0 to <35.0 kg/m2.
4. Able to comply with the time requirements for study visits and assessments.
5. Currently on cART for at least 24 months with two consecutive plasma HIV-1 RNA < 50 copies/ml at least 12 months apart.
6. CD4+ T-cell count ≥ 250 cells/µl (including borderline values) and CD4/CD8 < 0.9 during the screening period.
7. Agree to adhere to contraception during participation in the project and for 6 months after completion of the trial.
8. Willing to sign the informed consent form.

Exclusion Criteria:

1. Subjects who have had any serious acute illness within 8 weeks.
2. Subjects with a history of active autoimmune disease or autoimmune disease requiring systemic therapy.
3. Pre-treatment/exposure to any other immune checkpoint inhibitors [e.g., anti-programmed cell death protein 1 (PD-1), anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.].
4. The patient has been treated with

   1. Received previous treatment with other anti-submarine drugs within 30 days prior to enrollment.
   2. Received radiotherapy or chemotherapy 30 days prior to screening.
   3. Received immunosuppressive therapy 60 days prior to screening.
   4. Treatment with immunomodulators (e.g., interleukins, interferons), hydroxyurea, or phosphonates 60 days prior to screening.
   5. HIV vaccine or systemic cytotoxic chemotherapy 60 days prior to screening.
   6. Prior immunoglobulin (IgG) therapy.
   7. Previous blood transfusion or cell growth factor therapy 90 days prior to screening.
   8. Use of rifampicin, rifabutin, etc. at the time of screening or during the planned treatment phase.
5. Laboratory tests meet the following criteria.

   1. absolute neutrophil count (ANC) <1.50×109/L; hemoglobin (Hb) <105 g/L (male) or <95 g/L (female); platelets <75×10^9/μ L; international normalized ratio (INR) >1× upper limit of normal (ULN).
   2. Serum alanine aminotransferase (SGPT/ALT) >1.5× upper limit of normal (ULN), serum aspartate aminotransferase (SGOT/AST) >1.5× upper limit of normal (ULN), total bilirubin, direct bilirubin >1.5× upper limit of normal (ULN), serum creatinine >1.5× upper limit of normal (ULN) × upper limit of normal value (ULN).
   3. Five abnormal thyroid functions with clinical significance: tests include triiodothyronine (T3), tetraiodothyronine (T4), free triiodothyronine (FT3), free tetraiodothyronine (FT3), free tetraiodothyronine (FT4), and thyroid stimulating hormone (TSH).
   4. Abnormal and clinically significant adrenaline tests, which must include at least ACTH and cortisol. Abnormal and clinically significant blood glucose and glycated hemoglobin.
6. Abnormal and clinically significant twelve-lead ECG at the time of enrollment.
7. Subjects with interstitial changes on chest CT at the time of enrollment.
8. Subjects with severe cardiac disease, symptomatic or asymptomatic arrhythmias.
9. Patients with co-infection with HBV, HCV, syphilis, etc., patients with diabetes mellitus, and patients with other liver diseases.
10. Subjects with a history of active or suspected malignancy or malignant disease (except basal cell skin cancer or in situ cervical cancer) within five years.
11. Subjects with a history of tuberculosis or active tuberculosis.
12. Subjects with psychiatric or substance abuse disorders known to interfere with study requirements.
13. Subjects who have received immunomodulation or immunosuppression within 24 weeks prior to the first dose of study drug (including any dose of IV/oral [PO] steroids, but excluding steroids by inhalation, topical, or by local injection) within 24 weeks prior to the first dose of the study drug.
14. Pregnant and lactating women, or men and women who intend to conceive a child during the study period.
15. Psychiatric patients or those whose substance abuse interferes with the conduct of the trial.
16. Histone deacetylase inhibitors, such as valproate, butyrate, and phenylbutyrate, but may be enrolled after a 28-day elution period.
17. Patients with severe cardiac insufficiency [New York Heart Association (NYHA) Cardiac Insufficiency Classification Class IV].
18. Any arterial thromboembolic event, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, within 6 months prior to enrollment; normatively treated uncontrolled hypertension (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg); cardiomyopathy
19. Patients with significant QT/QTC interval during the screening period (Fridericia formula.

(19) Patients with a significant prolongation of the QT/QTC interval (Fridericia formula: QTcF=QT/RR0.33) during the screening period (e.g., repeated measurements showing a QTc interval >450 ms, or another risk of torsional ventricular tachycardia [TdP] [e.g., heart failure, hypokalemia, familial long QT syndrome]) or combination of drugs that may cause prolongation of the QT/QTc interval.

(20) Known allergy or anti-drug antibodies to drugs or excipients used in this trial.

(21) Those who are judged by the investigator to be unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
HIV-1 DNA levels | 52 weeks
  Change in HIV-1 DNA levels from baseline at each cycle of treatment

SECONDARY OUTCOMES:
CD4+ T-cell count, CD4+ T-cell percentage, CD8+ T-cell count, CD4+/CD8+ ratio | 52 weeks
  Changes in CD4+ T-cell count, CD4+ T-cell percentage, CD8+ T-cell count, CD4+/CD8+ ratio, and change from baseline at each cycle of treatment
HIV gag-specific CD8+ T ratio | 52 weeks
  Change from baseline in HIV gag-specific CD8+ T ratio at each cycle of treatment
HIV-1 RNA | 52 weeks
  Change in HIV-1 RNA from baseline at each cycle of treatment

OTHER OUTCOMES:
Treatment-Emergent Adverse Events | 52 weeks
  All adverse events occurred after drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu L, Zheng Z, Xun J, Liu L, Wang J, Zhang X, Shao Y, Shen Y, Zhang R, Zhang M, Sun M, Qi T, Wang Z, Xu S, Song W, Tang Y, Zhao B, Song Z, Routy JP, Lu H, Chen J. Anti-PD-L1 antibody ASC22 in combination with a histone deacetylase inhibitor chidamide as a "shock and kill" strategy for ART-free virological control: a phase II single-arm study. Signal Transduct Target Ther. 2024 Sep 9;9(1):231. doi: 10.1038/s41392-024-01943-9. PMID 39245675